CLINICAL TRIAL: NCT04773080
Title: Incidence, Risk Factors and Consequences of Acute Kidney Injury in Patients Undergoing Esophageal Cancer Surgery: a Historical Cohort Study
Brief Title: Incidence, Risk Factors and Consequences of Acute Kidney Injury in Patients Undergoing Esophageal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Ilaria Godi, Principal Investigator, Azienda Ospedaliera di Padova
Other Study IDs: 3073
Record Dates: First submitted 2021-01-25; First posted 2021-02-26 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Acute Kidney Injury; Postoperative Complications
MeSH Terms: conditions — Acute Kidney Injury; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- esophageal cancer surgery: patients undergoing elective esophageal surgery for cancer

SUMMARY:
Esophagectomy serves as an exemplar of major operative trauma, with well-known risk of pulmonary, cardiac, anastomotic, and septic complications and the presence of postoperative complications after esophagectomies for cancer is associated with a reduced long-term survival. There is a paucity in the literature regarding postoperative renal outcomes after esophageal surgery, with a wide range of incidence.

The investigators will conduct a historical cohort study aiming to evaluate the incidence of postoperative acute kidney injury in patients undergoing elective esophageal cancer surgery. Secondary, the investigators will assess the progression of the acute injury and the association with adverse pulmonary, cardiac, anastomotic, and septic events, as well as increase in hospital stay and mortality. The investigators will also identify risk factors associated with acute kidney injury occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Elective esophagectomy

Exclusion Criteria:

* End-stage renal disease
* Missing data for acute kidney injury definition
* Second surgery (for patients having multiple surgeries performed during a 30-day period, only the first in each period will be included)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent elective esophageal surgery for cancer
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative acute kidney injury | within 48 hours after surgery
  according to KDIGO criteria

SECONDARY OUTCOMES:
Incidence of transient or persistent postoperative acute kidney injury | 48 hours after development of acute kidney injury
  according KDIGO criteria
Number of patients with renal recovery | at 7 days, after 30 days and 3 months
  according ADQI criteria
Incidence of postoperative pulmonary complications | within 30 days after surgery
  based on European Perioperative Clinical Outcome (EPCO) definitions
Incidence of major adverse cardiac and cerebrovascular events (MACCE) | within 30 days after surgery
  composite outcome of non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure, new cardiac arrhythmia, angina, ischemic stroke
Incidence of sepsis | within 30 days after surgery
  according Sepsis-3 definition
Mortality in hospital | 1 year
  any death during the admission when the operation was performed
Increase in length of hospital stay | 1 year
  compared to the expected length of hospital stay according ACS NSQIP calculation

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Godi, MD, Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT04773080/Prot_SAP_000.pdf